CLINICAL TRIAL: NCT04573036
Title: A Phase 1, Single Center, Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and the Effect of Food on the Pharmacokinetics of HRS4800 in Healthy Male Participants
Brief Title: A Trial of HRS4800 Tables in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Atridia Pty Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HRS4800-I-101-AUS
Record Dates: First submitted 2020-09-16; First posted 2020-10-05 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-07

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Intervention Model Description: The study consists of 2 parts: single dose escalation (Part 1) with four cohorts and food effect on HRS4800 PK (Part 2) with one cohort. All cohorts can enroll healthy male subjects
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HRS4800 tablets cohort 1 (Experimental): Part 1 - HRS4800 Single Ascending Dose
  Interventions: Drug: HRS4800 tablets
- HRS4800 tablets cohort 2 (Experimental): Part 1 - HRS4800 Single Ascending Dose
  Interventions: Drug: HRS4800 tablets
- HRS4800 tablets cohort 3 (Experimental): Part 1 - HRS4800 Single Ascending Dose
  Interventions: Drug: HRS4800 tablets
- HRS4800 tablets cohort 4 (Experimental): Part 1 - HRS4800 Single Ascending Dose
  Interventions: Drug: HRS4800 tablets
- HRS4800 tablets cohort 5 (Experimental): Part 2 - HRS4800 Food Effect
  Interventions: Drug: HRS4800 tablets
- Placebo tablets (Placebo Comparator)
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: HRS4800 tablets — single oral administration
  Arms: HRS4800 tablets cohort 1; HRS4800 tablets cohort 2; HRS4800 tablets cohort 3; HRS4800 tablets cohort 4; HRS4800 tablets cohort 5
Drug: Placebo tablets — single oral administration
  Arms: Placebo tablets

SUMMARY:
This is a single-site study to evaluate the safety, tolerability and pharmacokinetics (PK) of single dose administration of HRS4800, and the effect of food on the PK of HRS4800 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the purposes and risks of the trial and comply with all study procedures before entering the trial, and provide signed informed consent.
* Male aged between 18 years and 55 years at screening, inclusive.
* Total body weight ≥50 kg at screening, and body mass index (BMI) between 18.0 and 32.0 kg/m2, inclusive.
* Agree to practice true abstinence; be surgically sterilised (performed at least 6 months prior and documented to no longer produce sperm - verbal confirmation through medical history review acceptable); or agree to use a condom if sexually active with a female partner of childbearing potential for at least 3 months after dosing.
* No clinically significant abnormalities in medical history, general physical examination, vital signs, laboratory tests (hematology, urinalysis, blood chemistry, coagulation function), and ECG, as determined by the investigator. Male aged between 18 years and 55 years at screening, inclusive.

Exclusion Criteria:

* History of severe digestive system disease or having a digestive disease currently within a month of screening or before first dosing, and may affect drug absorption or have safety risks.
* Severe infections, injuries or surgeries within 3 months of screening or before first dosing, or plan to undergo any surgeries during the trial.
* Use of any medicine affecting liver metabolism within 1 month of screening (see Appendix 1); use of any prescription medications within 14 days or 5 half-lives prior to dosing, use of any over-the-counter medicine or herbal products within 7 days prior to dosing; intention to use any other medicine during the trial.
* Whole blood donation or loss of more than 200 mL of blood within 1 month prior to dosing; or blood donation or loss of more than 400 mL of blood within 3 months prior to dosing; or plasma donation within 14 days prior to dosing; or received blood within 8 weeks prior to dosing.
* History of allergy to the study drug or any component of it.
* History of regular alcohol consumption in the past 1 month exceeding an average weekly intake of 21 standard drinks: 1 drink=5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor).
* Subject has used more than 5 tobacco or nicotine-containing products per day in the 6 months prior to dosing and is unable to refrain from use of such products from at least 48 hours prior to check-in through to the final study visit.
* Treatment with an investigational drug within 30 days (or 5 half-lives, whichever is longer) of dosing.
* History of drug abuse within 2 years prior to screening.
* Other conditions or laboratory abnormality that may increase the risk associated with study participation or IP administration or interfere with the interpretation of study results and, at the discretion of the investigator, makes the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Part 1 - HRS4800 Single Dose Escalation - Safety | 14 days
  • Safety: Incidence and severity of adverse events (AEs), vital signs (pulse rate, respiratory rate, blood pressure, body temperature), physical examination, laboratory tests, electrocardiogram (ECG), etc.
Part 2 - HRS4800 Food Effect | 21 days
  • PK parameters of HRS4800 and its active drug SHR175593 in plasma: AUC0-t
Part 2 - HRS4800 Food Effect | 21 days
  • PK parameters of HRS4800 and its active drug SHR175593 in plasma: AUC0-∞
Part 2 - HRS4800 Food Effect | 21 days
  • PK parameters of HRS4800 and its active drug SHR175593 in plasma: Tmax、
Part 2 - HRS4800 Food Effect | 21 days
  • PK parameters of HRS4800 and its active drug SHR175593 in plasma: Cmax
Part 2 - HRS4800 Food Effect | 21 days
  • PK parameters of HRS4800 and its active drug SHR175593 in plasma: t1/2、CL/F、Vz/F.

SECONDARY OUTCOMES:
Part 1 - HRS4800 Single Dose Escalation - PK | 14 days
  • PK parameters of HRS4800 and its active drug SHR175593 in plasma: AUC0-t
Part 1 - HRS4800 Single Dose Escalation - PK | 14 days
  AUC0-∞、
Part 1 - HRS4800 Single Dose Escalation - PK | 14 days
  Tmax
Part 1 - HRS4800 Single Dose Escalation - PK | 14 days
  Cmax
Part 1 - HRS4800 Single Dose Escalation - PK | 14 days
  t1/2
Part 1 - HRS4800 Single Dose Escalation - PK | 14 days
  CL/F、Vz/F.

CONTACTS AND LOCATIONS:
Overall Officials: Na Li, Study Director — Jiangsu Hengrui Pharmaceutical Co., Ltd.
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia